CLINICAL TRIAL: NCT05061758
Title: A Phase 2 Double Blind, Randomized, Placebo Controlled Trial inVEstigating the Effect and Safety of Several Dosing Regimens of LY3056480 in Patients With STAble Sensorineural Hearing Loss
Brief Title: A Trial of LY3056480 in Patients With SNLH
Acronym: VESTA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study put on hold
Sponsor: Audion Therapeutics BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUT-003
Record Dates: First submitted 2021-09-15; First posted 2021-09-30 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: double blinded, randomized, placebo controlled, multi center efficacy phase 2 study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Four injections of 250µg LY3056480 (Experimental): The treatment will be given transtympanically over the course of 2-7 weeks, according to dosing regimens below.
  * Group 1 - Regimen 1. Day 1, Day 4, Day 8, Day 11
  * Group 2 - Regimen 2. Weekly
  * Group 3 - Regimen 3. Every two weeks
  Interventions: Drug: LY3056480
- Four injections of placebo (Placebo Comparator): The treatment will be given transtympanically over the course of 2-7 weeks, according to dosing regimens below.
  * Group 1 - Regimen 1. Day 1, Day 4, Day 8, Day 11
  * Group 2 - Regimen 2. Weekly
  * Group 3 - Regimen 3. Every two weeks
  Interventions: Drug: LY3056480

INTERVENTIONS:
Drug: LY3056480 — LY3056480 is an inhibitor of gamma-secretase

SUMMARY:
A phase 2 trial with LY3056480 in patients with stable SNHL

DETAILED DESCRIPTION:
VESTA is a double blinded, randomized, placebo controlled, multi center efficacy phase 2 study comparing three dosing regimens of 250 µg LY3056480. Adult volunteers with stable mild to moderately-severe SNHL will be recruited through Adult Otolaryngology - Head & Neck Surgery Services in the US. Four injections of 250µg LY3056480 or placebo administered trans-tympanically into one ear (worse hearing ear).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 - 65 years of age;
2. Minimum of six months of documented stable hearing loss (+/- 5dB);
3. A documented stable word recognition test (stable for ~ 6 months +/- 6%/3 words)

Exclusion Criteria:

1. Presenting with a primary complaint of tinnitus
2. Any conductive hearing loss of greater than 15 dB at a single frequency or greater than 10 dB at two or more contiguous octave frequencies in the study ear
3. History of suspected or diagnosed genetic cause of hearing loss;
4. Partial deafness as defined as hearing loss in any frequency (up to 8 kHz) greater than 80dB
5. Suspected or known diagnosis of the following inner ear pathology, congenital hearing loss, fluctuating hearing loss, Ménière's disease, or secondary endolymphatic hydrops, perilymph fistula, cochlear barotrauma, autoimmune hearing loss, radiation-induced hearing loss, retro-cochlear lesion, ototoxicity
6. Evidence of acute or chronic otitis media or otitis externa on examination; or a history of middle ear pathology and/or surgery (except for ear tubes as a child)
7. Any therapy known as ototoxic
8. Participant in a previous trial of LY3056480

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
the efficacy of local treatment with LY3056480 in terms of hearing function | 6 months
  • Number of drug responders with at least a 2dB improvement in an adaptive sentence in noise test (international matrix test) compared to placebo

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - New York Eye and Ear Infirmary ICAHN school of Medicine Mount Sinai, New York, New York
  - Eastern Virginia Medical School, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Undecided